CLINICAL TRIAL: NCT03011970
Title: Temporal Dynamics and Pharmacokinetics of Intranasally Administered Oxytocin
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Bonn (Other)
Responsible Party: Principal Investigator, Rene Hurlemann, Professor, University Hospital, Bonn
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Basic Science
Other Study IDs: OXT_KINO
Record Dates: First submitted 2016-12-12; First posted 2017-01-06 (Estimated); Last update posted 2017-01-06 (Estimated); Status verified 2017-01

CONDITIONS: Healthy
MeSH Terms: interventions — Oxytocin

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Oxytocin; 24IU, 15min (Active Comparator): Intranasal administration, 24 international units (IU) oxytocin. Imaging starting 15min after nasal spray administration.
  Interventions: Drug: Oxytocin
- Oxytocin; 24IU, 45min (Active Comparator): Intranasal administration, 24 IU oxytocin. Imaging starting 45min after nasal spray administration.
  Interventions: Drug: Oxytocin
- Oxytocin; 24IU, 75min (Active Comparator): Intranasal administration, 24 IU oxytocin. Imaging starting 75min after nasal spray administration.
  Interventions: Drug: Oxytocin
- Oxytocin; 12IU, 45min (Active Comparator): Intranasal administration, 12 IU oxytocin. Imaging starting 45min after nasal spray administration
  Interventions: Drug: Oxytocin
- Oxytocin; 48IU, 45min (Active Comparator): Intranasal administration, 48 IU oxytocin. Imaging starting 45min after nasal spray administration
  Interventions: Drug: Oxytocin
- Placebo (Placebo Comparator): Placebo nasal spray.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oxytocin
  Arms: Oxytocin; 12IU, 45min; Oxytocin; 24IU, 15min; Oxytocin; 24IU, 45min; Oxytocin; 24IU, 75min; Oxytocin; 48IU, 45min
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether effects of intranasal oxytocin on amygdala response vary as a function of treatment dose and dose-test latency.

DETAILED DESCRIPTION:
The objective of the present study is to determine whether intranasal oxytocin (IN-OXT) effects on blood oxygenation level-dependent functional magnetic resonance imaging (BOLD fMRI) in the amygdala vary as a function of dose and latency. In particular, the investigators plan to compare effects of three different IN-OXT doses (12, 24, and 48 international units, IU) and three different dose-test latencies of IN-OXT administration (task starting at 15, 45 and 75min after administration) on established neural and behavioural correlates of emotion processing. As effects of OXT are particularly promising in autism, the investigators further want to investigate how autistic-like traits influence the OXT effects in exploratory post-hoc analyses

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers
* Right-handed

Exclusion Criteria:

* Current or past psychiatric disease
* Current or past physical illness
* Psychoactive medication
* Tobacco smokers
* MRI contraindication (e.g. metal in body, claustrophobia)

Ages: 18 Years to 40 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 116 (Actual)
Dates: Start 2014-09; Primary Completion 2015-12 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Neural substrates of emotion processing, measured via blood-oxygen-level dependent signal in the amygdala | 45min after nasal spray administration
  Magnetic resonance imaging (MRI) will be performed to measure blood-oxygen-level dependent signal in response to emotional face stimuli of varying intensity. The investigators specifically plan to investigate amygdala response to fearful faces, as this subcortical region has repeatedly been reported to show activation changes after OXT treatment.
  Dose-test latency varies between the different treatment arms (i.e. imaging starts 15min [arm 1], 45min [arm 2,4 and 5] or 75min [arm 3] after nasal spray administration).

SECONDARY OUTCOMES:
Ratings of emotional faces | 45min after nasal spray administration
  During each trial, subjects are asked to use a button response grip to indicate whether they perceived the depicted face as neutral, fearful or happy.
  Depending on the treatment arm, ratings are recorded 15min (arm 1), 45min (arm 2,4 and 5) or 75min (arm 3) after nasal spray administration.
Questionnaire measurement of mood (PANAS) | 10 min before and 105 min after nasal spray administration
  Positive and negative affect is assessed via self-rating questionnaire 'The Positive and Negative Affect Schedule' using a categorical 5 point scale.
Questionnaire measurement of anxiety (STAI). | 10 min before and 105 min after nasal spray administration
  State anxiety is assessed via self-rating questionnaire 'and State Trait Anxiety Inventory' using a categorical 4 point scale.
Saliva oxytocin concentrations | immediately before the nasal spray administration and (on average) 15,40,80 and 105 min after administration
Plasma oxytocin concentrations | immediately before the nasal spray administration and immediately after the fMRI experiment
Modulatory effects of autistic like traits on neural and behavioral outcome measures | screening session, ~7days prior to imaging session
  Autistic like traits are assessed via Autism Spectrum quotient in a screening session, preceding the testing sessions. The investigators expect pronounced OXT effects in subjects with high autistic-like traits.

CONTACTS AND LOCATIONS:
Locations (1):
- Department of Psychiatry, University of Bonn, Bonn, North Rhine-Westphalia, Germany